CLINICAL TRIAL: NCT03820609
Title: Interactive Digital Intervention to Prevent Violence Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Happy People Games, LLC (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HappyPeopleGames
Record Dates: First submitted 2018-10-30; First posted 2019-01-29 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Sexual Assault
Keywords: Sexual Assault; Digital Intervention

STUDY DESIGN:
Intervention Model Description: A non-randomized open trial with a 1-month follow up will assess preliminary effects on attitudes and behaviors, and will establish procedures for assessing change in proximal (attitude) and distal (behavioral) outcomes in preparation for large-scale evaluation in a Phase 2 SBIR proposal.
Masking Description: The outcome evaluation is a non-randomized open pilot trial. Therefore, all participants and project collaborators are aware that individuals enrolled in the study are asked to complete the prevention program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Intervention (Experimental): Make a Change is a universal sexual assault (SA) prevention program that aligns with best-practices in prevention, utilizes the theory and strategies of serious games for health, and addresses risk and protective factors for SA across the social ecology of individual, peer and community factors that foster SA. This novel digital application also leverages theories of behavior change within serious games for health, and integrates successful practices in videogame design to promote engagement, learning and skill-building.
  Interventions: Behavioral: Digital Intervention

INTERVENTIONS:
Behavioral: Digital Intervention — This digital application for sexual assault prevention can be completed on a tablet computer.

SUMMARY:
The primary aim of this Phase I SBIR is to create and test an alpha version of Make a Change for mobile devices, and to document the technical merit, commercial viability, and proof of concept of the product. Successful completion of this proposal will result in the creation of two assets: 1) an "Intervention Manual" that (similar to a logic model) will align key game mechanics with theory and behavior change goals and, 2) the digital application for mobile devices. Focus groups and interviews with students, as well as interviews with campus stakeholders, will be used to inform development of the digital application and ensure its commercial viability. A non-randomized open trial with a 1-month follow up will assess preliminary effects on attitudes and behaviors, and will establish procedures for assessing change in proximal (attitude) and distal (behavioral) outcomes in preparation for large-scale evaluation in a Phase 2 SBIR proposal. This line of research and development has the potential to develop a commercially viable product with high public health impact that can be disseminated to 1700+ community colleges and 3,000+ 4-year colleges, and readily adapted to high schools, clinics and military settings.

DETAILED DESCRIPTION:
Sexual assault (SA) is prevalent among students at 2- and 4-year colleges. The rate of SA among college students is three times greater than the rate in the general population, making prevention on college campuses a public health priority. There are no college SA prevention programs that document reductions in SA in a rigorous research design. Digital applications that use the theory and strategies of serious games integrate proven theories of behavior change (social cognitive theory, self-determination theory) to produce sustained, measurable behavioral outcomes, and are effective for promoting change in a range of health behaviors. Digital applications have high market potential in light of widespread use of mobile devices among young adults. Problematically, there are no commercially-available digital applications for SA prevention with efficacy in reducing SA. Accordingly, in this proposal, the Interactive Digital Intervention to Prevent Violence among Young Adults team will design, create and pilot the Make a Change digital application. Make a Change is a universal prevention program that aligns with best-practices in prevention, utilizes the theory and strategies of serious games for health, and addresses risk and protective factors for SA across the social ecology of individual, peer and community factors that foster SA. This novel digital application also leverages theories of behavior change within serious games for health, and integrates successful practices in videogame design to promote engagement, learning and skill-building. This team consists of experts in SA prevention, commercial videogame production, the development and testing of serious games for health, and business development and marketing. The primary aim of this Phase I SBIR is to create and test an alpha version of Make a Change for mobile devices, and to document the technical merit, commercial viability, and proof of concept of the product. Successful completion of this proposal will result in the creation of two assets: 1) an "Intervention Manual" that (similar to a logic model) will align key game mechanics with theory and behavior change goals and, 2) the digital application for mobile devices. Focus groups and interviews with students, as well as interviews with campus stakeholders, will be used to inform development of the digital application and ensure its commercial viability. A non-randomized open trial with a 1-month follow up will assess preliminary effects on attitudes and behaviors, and will establish procedures for assessing change in proximal (attitude) and distal (behavioral) outcomes in preparation for large-scale evaluation in a Phase 2 SBIR proposal. This line of research and development has the potential to develop a commercially viable product with high public health impact that can be disseminated to 1700+ community colleges and 3,000+ 4-year colleges, and readily adapted to high schools, clinics and military settings.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 24
* Enrolled as a student at one of the study sites

Exclusion Criteria:

* None

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Sexual aggression | 1-month follow-up
  Assessed via the Sexual Experiences Survey - Revised
Sexual victimization | 1-month follow-up
  Assessed via the Sexual Experiences Survey - Revised
Bystander intervention | 1-month follow-up
  Assessed via the Bystander Attitudes Survey

SECONDARY OUTCOMES:
Rape supportive beliefs | 1-month follow-up
  Assessed via the Short-Form Illinois Rape Myth Acceptance Scale
Perception of peer support for sexual aggression | 1-month follow-up
  Assess through items from Boeringer's Social Norms Measure and Clemson's Peer Pressure Measure
Perceived peer norms | 1-month follow-up
  Change in the accuracy in perception of peer norms (assessed via responses to in-app questions)
Bystander intervention confidence | 1-month follow-up
  Assessed via the Bystander Efficacy Scale from ARC-3
Communication of consent | 1-month follow-up
  Assessed via the Consent Experiences Scale
Self-protective behavior | 1-month follow-up
  Assessed via the Alcohol Use Self-Protective Behavior Scale
Psychological barriers to resistance | 1-month follow-up
  Assessed via the Psychological Barriers to Resistance Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wood, Principal Investigator — Happy People Games
Locations (2):
- United States (2):
  - Community College of Rhode Island, Warwick, Rhode Island
  - Clemson University, Clemson, South Carolina

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan.